CLINICAL TRIAL: NCT02419391
Title: A Randomized, Single-blind, Placebo-controlled Phase I Trial to Evaluate the Safety, Tolerability and Immunogenicity of the Recombinant MVA BN® RSV Vaccine in Healthy Adult Subjects
Brief Title: Trial to Evaluate the Safety, Tolerability and Immunogenicity of the Recombinant MVA BN® RSV Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RSV-MVA-001
Record Dates: First submitted 2015-04-07; First posted 2015-04-17 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: RSV Vaccines; Respiratory Syncytial Virus Vaccines
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): 18-49 year old healthy subjects, receiving either 1x10E7TCID50 MVA BN RSV or Placebo
  Interventions: Biological: MVA BN RSV; Other: Placebo
- Group 2 (Experimental): 18-49 year old healthy subjects, receiving either 1x10E8TCID50 MVA BN RSV or Placebo
  Interventions: Biological: MVA BN RSV; Other: Placebo
- Group 3 (Experimental): 50-65 year old healthy subjects, receiving either 1x10E8TCID50 MVA BN RSV or Placebo
  Interventions: Biological: MVA BN RSV; Other: Placebo

INTERVENTIONS:
Biological: MVA BN RSV — Liquid frozen suspension of MVA-mBN294B
  Other Names: MVA-mBN294B
Other: Placebo — Tris Buffered Saline, sterile
  Other Names: TBS

SUMMARY:
A total of 63 subjects will be recruited into three groups (18 subjects per group will receive MVA BN RSV vaccine and three subjects per group will receive placebo). Liquid frozen suspension of MVA BN RSV.

Each subject will receive two vaccinations with either MVA-BN RSV vaccine 1 x 108 TCID50 per 0.5 ml, 1 x 107 TCID50 per 0.5 ml or with placebo.

ELIGIBILITY:
Inclusion Criteria:

* signed and dated an informed consent form
* Body mass index ≥ 18.5 and < 35.
* Women of childbearing potential (WOCBP) must have used an acceptable method of contraception

Exclusion Criteria:

* Pregnant or breast-feeding women.
* Uncontrolled serious infection, i.e. not responding to antimicrobial therapy.
* History of any serious medical condition.
* History of or active autoimmune disease.
* Known or suspected impairment of immunologic functions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2015-08; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Occurrence of serious adverse events | Screening up to week 34 after first vaccination
  Occurrence, relationship to the trial vaccine and intensity of any serious adverse event (SAE).
Occurrence of grade 3 adverse events | Screening up to week 8 after first vaccination
  Occurrence of any grade 3 or higher adverse events possibly, probably or definitely related to the trial vaccine within four weeks after each vaccination.
Solicited local adverse events | day of vaccination and the following seven days
  Occurrence, intensity and duration of solicited local adverse events after each vaccination Occurrence, intensity and duration of solicited local adverse events after each vaccination Occurrence, intensity and duration of solicited local adverse events after each vaccination
Unsolicited non-serious adverse events | within four weeks after each vaccination
  Occurrence, relationship to the trial vaccine and intensity of unsolicited non-serious adverse events
Solicited general adverse events | day of vaccination and the following seven days
  Occurrence, relationship to the trial vaccine, intensity and duration of solicited general adverse events

SECONDARY OUTCOMES:
Vaccinia-specific cellular immune responses. | cellular immune response measured up to week 4 after 2nd vaccination
  To assess the RSV-specific and vaccinia-specific cellular immune responses against the MVA-BN RSV vaccine in healthy adult subjects. Spot forming units will be determined by using an IFN-γ ELISPOT assay.
RSV-specific humoral immune response | humoral immune response is measured up to week 34
  To assess the RSV-specific serum antibody responses by ELISA
RSV-specific humoral immune response | humoral immune response is measured up to week 34
  To assess the RSV-specific serum antibody responses by PRNT
RSV-specific humoral immune response | humoral immune response is measured up to week 34
  To assess the RSV-specific mucosal antibody responses by ELISA
Vaccinica-specific humoral immune response | humoral immune response is measured up to week 34
  To assess the Vaccinica-specific serum antibody responses by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Casey Johnson, DO, Principal Investigator — Johnson County Clin-Trials (JCCT)
Locations (1):
- Johnson County Clin-Trials (JCCT), Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided